CLINICAL TRIAL: NCT05456958
Title: Self-regulation of Post-traumatic Stress Disorder (PTSD) Neurocircuitry Using Multiple Sessions of Real-Time Functional Magnetic Resonance Imaging (RtfMRI)
Brief Title: Multi-session fMRI-Neurofeedback in PTSD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Nicholson (Other)
Collaborators: McMaster University (Other); University of Ottawa (Other); Western University (Other)
Responsible Party: Sponsor-Investigator, Andrew Nicholson, Adjunct Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANicho01
Record Dates: First submitted 2022-06-30; First posted 2022-07-13 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Real-time neurofeedback; Functional magnetic resonance imaging (fMRI); Post-traumatic stress disorder (PTSD); Posterior cingulate cortex (PCC); Amygdala
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: PTSD participants (N=60) will be randomly assigned to receive neurofeedback targeting one of two regions-of-interest - amygdala (N=20) or PCC (N=20) - or to the sham-control arm (N=20), where individuals will receive a fake neurofeedback signal (i.e., from a successful participant in one of the experimental arms, thereby controlling for motivational effects).
Who Masked: Participant, Investigator
Masking Description: Both investigators and participants will be blinded with regards to arm assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Amygdala (Experimental): PTSD participants will receive a neurofeedback signal reflecting amygdala activity.
  Interventions: Other: MRI Biofeedback
- Posterior cingulate cortex (PCC) (Experimental): PTSD participants will receive a neurofeedback signal reflecting PCC activity.
  Interventions: Other: MRI Biofeedback
- Sham-control (Experimental): PTSD participants will receive a sham neurofeedback signal, i.e., from a successful participant in one of the experimental arms.
  Interventions: Other: Sham-MRI Biofeedback

INTERVENTIONS:
Other: MRI Biofeedback — We will use state-of-the-art fMRI and neurofeedback of brain signals in order to teach patients with PTSD to self-regulate pathological brain activity that is associated with their symptoms. Indeed, feedback information is crucial for learning, where rt-fMRI-based neurofeedback makes information about brain activity accessible to our consciousness (Ros et al., 2014; Sitaram et al., 2017). It thus provides a reinforcement signal to induce personalized learning mechanisms, allowing individuals to search for appropriate cognitive strategies to voluntarily control brain activity. The feedback signal will come from activity within either the amygdala or PCC.
  Arms: Amygdala; Posterior cingulate cortex (PCC)
Other: Sham-MRI Biofeedback — In the sham-control arm (N=20), individuals will receive fake neurofeedback signal, i.e., from a successful participant in one of the experimental arms.
  Arms: Sham-control

SUMMARY:
Post-traumatic stress disorder (PTSD) is a debilitating and highly prevalent psychiatric disorder that develops in the aftermath of trauma exposure (APA, 2013). PTSD has been strongly associated with altered activation patterns within several large-scale brain networks and, as such, it has been suggested that normalizing pathological brain activation may be an effective treatment approach.

The objective of this proposed study is to investigate the ability of PTSD patients to self-regulate aberrant neural circuitry associated with PTSD psychopathology using real-time functional magnetic resonance imaging (rt-fMRI) neurofeedback. Here, the investigators are building upon previous single-session pilot studies examining the regulation of the amygdala and the posterior cingulate cortex (PCC) in PTSD (Nicholson et al., 2021) (Nicholson et al., 2016) by: (1) Examining the effect of multiple sessions of rt-fMRI neurofeedback and, (2) Comparing PCC- and amygdala-targeted rt-fMRI neurofeedback to sham-control groups with regards to changes in PTSD symptoms and neural connectivity.

DETAILED DESCRIPTION:
Overview of Study Procedure:

This study consists of the following components:

1. Clinical assessment
2. 5 x self-report symptom assessment battery that will be administered electronically via REDCap (Research Electronic Data Capture), a secure web application for building and managing online surveys and databases.
3. 3 x rt-fMRI neurofeedback sessions, plus a 30-minute semi-structured qualitative interview immediately after the end of scanning with a trauma-informed and clinically trained graduate student
4. 7 weeks of actigraphy device usage to monitor participant biological (sleep) rhythms and physical activity.

(1) Clinical Assessment: Those who meet criteria for inclusion will be scheduled for baseline clinical assessments. Baseline clinical assessments will include the Mini-International Neuropsychiatric Interview (MINI; (Sheehan et al., 1998), and the Clinician-Administered PTSD Scale-5 (CAPS-5; (Weathers et al., 2018). The MINI will be used to establish mental health disorder diagnoses, and the CAPS will be used to establish a primary diagnosis of PTSD and symptom severity. In keeping with previous single-session studies by our group (Nicholson et al., 2016; 2021), during the clinical assessment session PTSD participants will be asked to select personalized trauma-associated words that induce emotional responses as well as neutral words associated with neutrally salient memories. The chosen words will be utilized for the emotion induction paradigm during neurofeedback. To ensure that the words only induce moderate emotional arousal, participants will self-report levels of distress associated with viewing the words and selection will be limited to words with a maximum distress rating of 7/10.

(2) Self-report Assessments (via REDCap): In this study, participants will also complete a battery of self-report questionnaires prior to the first neurofeedback session, including: Life Events Checklist (LEC-5) (Weathers et al., 2013), Beck Depression Inventory (BDI) (Beck et al., 1997), Childhood Trauma Questionnaire (CTQ) (Bernstein et al., 2003), Difficulties in Emotion Regulation Scale (DERS) (Perasso & Velotti, 2017), Multiscale Dissociation Inventory (MDI) (Briere et al., 2005), the Depression Anxiety Stress Scale-21 (DASS-21) (Lovibond & Lovibond, 1995), the Multidimensional Assessment of Interoceptive Awareness (MAIA) (Mehling et al., 2012), the Insomnia Severity Index (ISI) (Morin et al., 2011), and the PTSD Checklist for DSM-5 (PCL-5) (Blevins et al., 2015). The PCL-5, BDI, DERS, MDI, DASS-21, ISI, and MAIA will be completed again after each rt-fMRI session, as well as at a 1- month follow-up. This battery of questionnaires will be administered at each time interval via REDCap.

(3) rt-fMRI Neurofeedback Sessions: In this study, the investigators will employ a 3 arm (amygdala vs. PCC vs. sham-control) vs 3 session design. fMRI data will be acquired using a 3T whole-body MRI scanner at St. Joseph's Hospital, London, Ontario, which is associated with the University of Western Ontario. All participants will undergo 3 rt-fMRI training sessions over the course of a 3-week period (1 session per week). fMRI data will be acquired using a 3T whole-body MRI scanner (Magnetom Tim Trio, Siemens Medical Solutions, Erlangen, Germany), equipped with a 32-channel phased array head coil.

rt-fMRI sessions: At the start of each session and after each run within a session, participants will also be asked to measure their state PTSD and dissociative symptoms using the Response to Script-Driven Imagery Scale (RSDI). The RSDI is a brief, self-report, 7-item Likert scale (Hopper et al 2007) and will be administered to participants while they are inside the scanner. Each rt-fMRI session will proceed as follows: a pre-session RSDI, a localization scan, an anatomical scan, an initial resting-state scan, 4 task runs (~8 minutes per run; with an RSDI after each task run), followed by another resting-state scan. For each rt-fMRI session, there will be 3 training runs, followed by a transfer run (to assess neurofeedback learning effects), for a total of 4 task runs. The transfer run is identical to the training runs except for the fact that participants will not receive any neurofeedback signal. The tasks and timing for all 3 rt-fMRI sessions will be identical.

rt-fMRI task: During the rt-fMRI task, the neurofeedback signal will based on participant's activity within either the PCC or amygdala, as per their randomized group assignment. Participants will be told that they will be "regulating brain activity in an area related to emotion." They will not be given any specific strategies with which to regulate brain activity, rather they will be advised to learn individualized strategies that work best for themselves in order to control the feedback signal. The task runs will consist of personalized trauma-associated words chosen by participants that induce emotional responses as well as neutral words. There are 3 different conditions that will occur during the task runs. Prior to each condition, participants will receive/read an instruction that will last approximately 2 seconds and indicates which condition will follow. In one third of the trials the condition will be 'regulate', during which participants will attempt to regulate their brain activity while viewing a trauma-associated word. In another one third of trials the condition will be 'view', during which participants will view a trauma-associated word without making any attempt to regulate their brain activity. In the final one third of the trials the condition will be 'neutral', during which participants will view a neutral word and not attempt to regulate brain activity. The order of the conditions within each task run will be counterbalanced. When presented, each word will be displayed for 24 seconds. Words will be presented using specialized fMRI stimulus delivery software (Presentation, Neurobehavioral Systems, Albany, CA, USA). Participants in the sham-control arm (N=20), will receive a fake neurofeedback signal (i.e., from a successful participant in one of the experimental arms, thereby controlling for motivational effects). Otherwise, the rt-fMRI task and all instructions provided will be identical for participants in the sham-control arm.

Neurofeedback task: During the presentation of words in the fMRI scanner, participants will be able to view a visual feedback display in the form of a thermometer-like bar graph. The number of bars displayed will reflect the amplitude increase of the fMRI signal in the region-of-interest (PCC or amygdala) relative to a baseline period. Feedback will occur every 2 seconds as represented by the number of changing bars. During the 'regulate' condition, participants will be asked to decrease the bars on the thermometer. During the 'view' and 'neutral' conditions, participants will be asked not to try to change the bars on the thermometer. Participants will not be given any specific strategies/guidance regarding how to regulate brain activity.

Qualitative interview: After completion of each fMRI scanning session, participants will complete a semi-structured qualitative interview with the investigator, outside of the scanner. The participants will be asked a number of questions regarding the cognitive strategies they employed to complete the task and their perceived efficacy of the various strategies used. As well, participants will be asked a number of questions relating to their subjective experiences (i.e., motivation, valence, frustration, mind-wandering, etc.) during neurofeedback training. The qualitative interviews will be recorded (via an audio recorder) and transcribed using a third-party transcription service. Any identifying information (i.e., participant name, affiliations, etc.) will be removed from the transcript so it is not possible to identify them from the interview. Transcripts from all participants will be 'pooled together' to analyze common themes across experiences.

(4) Actigraphy devices: Participants will wear a GENEActiv (Activinsights) actigraphy device throughout the duration of the study. The purpose of actigraphy measurements is to monitor participant biological (sleep) rhythms and physical activity. The GENEActive actigraphy device will be worn on the wrist and will collect continuous data at 30Hz.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Fluent English speaker
* Comfortable using electronic devices (i.e., laptop, tablet, smartphone, etc.)
* Meet criteria for a primary diagnosis of PTSD via the DSM-5 on the Clinician Administered PTSD Scale (CAPS-5). Note: given high rates of PTSD co-morbidity with major depressive disorder and anxiety disorders, these participants will not be excluded from the study, allowing for a naturalistic sample
* Able to provide written informed consent.

Exclusion Criteria:

Medical

* Pregnant women or women who are breastfeeding
* Serious illness (including cardiac, hepatic, renal, respiratory, endocrinologic, neurologic, or hematologic disease) that is not stabilized based on the judgment of primary investigator
* Contraindications for research MRI, including metallic implants
* Neurological disease, past head injury with loss of consciousness, stroke, seizures
* Major untreated medical illness (e.g., cancer, thyroid disorder)
* Any other condition that might interfere with the person's capacity to give informed consent, or to adhere to the study protocol.

Psychological/Psychiatric

* Active substance use or abuse as defined by the MINI or judged to be a problem by the PI
* Current or past pain disorders, bipolar disorders or psychosis, schizophrenia, and any other psychotic disorder will be excluded
* Participants will also be excluded for active suicidality, history of pervasive developmental disorders, or any other major medical illnesses
* Meeting criteria for substance use disorder in the past three months on the MINI
* Chronic opioid analgesic use within the last three months
* Any other condition that might interfere with the person's capacity to give informed consent, or to adhere to the study protocol
* Current engagement in a primary trauma-focused psychotherapy treatment.

Other

* History of claustrophobia
* Previous engagement in biofeedback, neurofeedback, or any form of brain stimulation therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants will be asked for both their biological sex and gender-identity on a demographic form at the start of the study.
Enrollment: 60 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Changes in PTSD symptoms over neurofeedback training sessions | Change in baseline (pre-neurofeedback) at 1-week intervals (i.e., post-neurofeedback session 1, 2, 3) and at a 1-month follow-up)
  The change in PTSD symptoms, as measured by PTSD Checklist 5 (PCL-5) scores, will be assessed over the course of 3 neurofeedback training sessions and at a 1-month follow-up. PCL-5 is a self-report measure used to gauge the DSM-5 symptoms of PTSD. PCL-5 scores range from 0 to 80 with higher scores indicating more severe PTSD symptoms.
Region-of-interest (ROI) downregulation analysis over neurofeedback training sessions | Change in ROI activation between neurofeedback sessions 1, 2, and 3
  In order to evaluate ROI downregulation (i.e., neurofeedback success), we will extract the event-related BOLD signal from the ROI during the regulate and view conditions.

SECONDARY OUTCOMES:
Change in depressive symptoms (i.e., BDI-II) over neurofeedback training sessions | Change in baseline (pre-neurofeedback) at 1-week intervals (i.e., post-neurofeedback session 1, 2, 3) and at a 1-month follow-up)
  The change in depressive symptoms will be assessed over the course of 3 neurofeedback training sessions and at a 1-month follow-up. Beck's Depression Inventory II (BDI-II) will be used to measure depressive symptoms. BDI-II scores range from 0 to 63 with higher scores indicating more severe depression symptoms.
Change in emotion regulation abilities (i.e., DERS) over neurofeedback training sessions | Change in baseline (pre-neurofeedback) at 1-week intervals (i.e., post-neurofeedback session 1, 2, 3) and at a 1-month follow-up)
  The change in emotion regulation abilities will be assessed over the course of 3 neurofeedback training sessions and at a 1-month follow-up. The Difficulties in Emotion Regulation (DERS) scale will be used to assess self-reported abilities in emotion regulation. DERS scores range from 36 to 180 with higher scores indicating greater problems with emotion regulation.
Change in trauma-related memory recall (i.e., RSDI) over neurofeedback training sessions | Change in baseline (pre-neurofeedback) at 1-week intervals (i.e., post-neurofeedback session 1, 2, 3) and at a 1-month follow-up)
  The change in trauma-related memory recall will be assessed over the course of 3 neurofeedback training sessions and at a 1-month follow-up. The Response to Script Driven Imagery (RSDI) scale will be used to assess trauma-related memory recall. RSDI scores range from 0 to 66 with higher scores indicating greater recall of trauma-related memories.
Change in dissociation symptoms (i.e., MDI) over neurofeedback training sessions | Change in baseline (pre-neurofeedback) at 1-week intervals (i.e., post-neurofeedback session 1, 2, 3) and at a 1-month follow-up)
  The change in dissociation symptoms will be assessed over the course of 3 neurofeedback training sessions and at a 1-month follow-up. The Multiscale Dissociation Inventory (MDI) scale will be used to assess PTSD-related dissociation symptoms. MDI scores range from 30 to 150 with higher scores indicating greater PTSD-related dissociation symptoms.
Change in emotional states of depression, anxiety, and stress (i.e., DASS-21) over neurofeedback training sessions | Change in baseline (pre-neurofeedback) at 1-week intervals (i.e., post-neurofeedback session 1, 2, 3) and at a 1-month follow-up)
  The change in emotional states of depression, anxiety, and stress symptoms will be assessed over the course of 3 neurofeedback training sessions and at a 1-month follow-up. The Depression, Anxiety and Stress Scale 21 (DASS-21) will be used to measure the PTSD-related emotional states of depression, anxiety, and stress. DASS-21 scores range from 0 to 63 with higher scores indicating greater depression, anxiety, and stress symptoms
Change in interoceptive awareness (i.e., MAIA) over neurofeedback training sessions | Change in baseline (pre-neurofeedback) at 1-week intervals (i.e., post-neurofeedback session 1, 2, 3) and at a 1-month follow-up)
  The change in interoceptive awareness will be assessed over the course of 3 neurofeedback training sessions and at a 1-month follow-up. The Multidimensional Assessment of Interoceptive Awareness (MAIA) will be used to assess interoceptive awareness. MAIA scores are averaged across items within 8 different sub-scales. Sub-scale average scores range from 0 to 5 with higher scores indicating greater interoceptive awareness.
Change in sleep difficulties (i.e., ISI) over neurofeedback training sessions | Change in baseline (pre-neurofeedback) at 1-week intervals (i.e., post-neurofeedback session 1, 2, 3) and at a 1-month follow-up)
  The change in sleep difficulties will be assessed over the course of 3 neurofeedback training sessions and at a 1-month follow-up. The Insomnia Severity Index (ISI) will be used to assess sleep difficulties. ISI scores range from 0 to 28 with higher scores indicating greater severity of insomnia.
Changes in biological (sleep) rhythms (i.e., actigraphy) over neurofeedback training sessions | Data collection will span 7-weeks during the study (i.e., 1-week baseline before neurofeedback session #1, 1-week between neurofeedback sessions #1 and #2, 1-week between neurofeedback sessions #2 and #3, 1-month follow-up after neurofeedback session #3)
  The change in biological (sleep) rhythms will be assessed over the course of 7-weeks during the study. The actigraphy devices will be used to assess biological (sleep) rhythms.
Changes in physical activity (i.e., actigraphy) over neurofeedback training sessions | Data collection will span 7-weeks during the study (i.e., 1-week baseline before neurofeedback session #1, 1-week between neurofeedback sessions #1 and #2, 1-week between neurofeedback sessions #2 and #3, 1-month follow-up after neurofeedback session #3)
  The change in physical activity will be assessed over the course of 7-weeks during the study. The actigraphy devices will be used to assess physical activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Lawson Health Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nicholson AA, Rabellino D, Densmore M, Frewen PA, Steryl D, Scharnowski F, Theberge J, Neufeld RWJ, Schmahl C, Jetly R, Lanius RA. Differential mechanisms of posterior cingulate cortex downregulation and symptom decreases in posttraumatic stress disorder and healthy individuals using real-time fMRI neurofeedback. Brain Behav. 2022 Jan;12(1):e2441. doi: 10.1002/brb3.2441. Epub 2021 Dec 18. PMID 34921746
- [Background] Nicholson AA, Rabellino D, Densmore M, Frewen PA, Paret C, Kluetsch R, Schmahl C, Theberge J, Neufeld RW, McKinnon MC, Reiss J, Jetly R, Lanius RA. The neurobiology of emotion regulation in posttraumatic stress disorder: Amygdala downregulation via real-time fMRI neurofeedback. Hum Brain Mapp. 2017 Jan;38(1):541-560. doi: 10.1002/hbm.23402. Epub 2016 Sep 20. PMID 27647695
- [Background] Weathers FW, Bovin MJ, Lee DJ, Sloan DM, Schnurr PP, Kaloupek DG, Keane TM, Marx BP. The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5): Development and initial psychometric evaluation in military veterans. Psychol Assess. 2018 Mar;30(3):383-395. doi: 10.1037/pas0000486. Epub 2017 May 11. PMID 28493729
- [Background] Weathers, F. W., Litz, B. T., Keane, T. M., Palmieri, P. A., Marx, B. P., & Schnurr, P. P. (2013). The ptsd checklist for dsm-5 (pcl-5). Scale available from the National Center for PTSD at www. ptsd. va. gov, 10(4), 206.
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Beck AT, Guth D, Steer RA, Ball R. Screening for major depression disorders in medical inpatients with the Beck Depression Inventory for Primary Care. Behav Res Ther. 1997 Aug;35(8):785-91. doi: 10.1016/s0005-7967(97)00025-9. PMID 9256522
- [Background] Bernstein DP, Stein JA, Newcomb MD, Walker E, Pogge D, Ahluvalia T, Stokes J, Handelsman L, Medrano M, Desmond D, Zule W. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. Child Abuse Negl. 2003 Feb;27(2):169-90. doi: 10.1016/s0145-2134(02)00541-0. PMID 12615092
- [Background] Perasso, Giulia & Velotti, Patrizia. (2017). Difficulties in Emotion Regulation Scale. 10.1007/978-3-319-28099-8_810-1.
- [Background] Briere J, Weathers FW, Runtz M. Is dissociation a multidimensional construct? Data from the Multiscale Dissociation Inventory. J Trauma Stress. 2005 Jun;18(3):221-31. doi: 10.1002/jts.20024. PMID 16281216
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Mehling WE, Price C, Daubenmier JJ, Acree M, Bartmess E, Stewart A. The Multidimensional Assessment of Interoceptive Awareness (MAIA). PLoS One. 2012;7(11):e48230. doi: 10.1371/journal.pone.0048230. Epub 2012 Nov 1. PMID 23133619
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Hopper, J. W., Frewen, P. A., Sack, M., Lanius, R. A., & van der Kolk, B. A. (2007). The responses to Script-Driven Imagery Scale (RSDI): Assessment of state posttraumatic symptoms for psychobiological and treatment research. Journal of Psychopathology and Behavioral Assessment, 29(4), 249-268. https://doi.org/10.1007/s10862-007-9046-0
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders (5th ed.). https://doi.org/10.1176/appi.books.9780890425596
- [Background] Ros T, J Baars B, Lanius RA, Vuilleumier P. Tuning pathological brain oscillations with neurofeedback: a systems neuroscience framework. Front Hum Neurosci. 2014 Dec 18;8:1008. doi: 10.3389/fnhum.2014.01008. eCollection 2014. PMID 25566028
- [Background] Sitaram R, Ros T, Stoeckel L, Haller S, Scharnowski F, Lewis-Peacock J, Weiskopf N, Blefari ML, Rana M, Oblak E, Birbaumer N, Sulzer J. Closed-loop brain training: the science of neurofeedback. Nat Rev Neurosci. 2017 Feb;18(2):86-100. doi: 10.1038/nrn.2016.164. Epub 2016 Dec 22. PMID 28003656
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Derived] Lieberman JM, Lanius RA, Theberge J, Frey BN, Frewen PA, Scharnowski F, Steyrl D, Ros T, Densmore M, Tassinari E, Matic V, Hosseini-Kamkar N, Narikuzhy S, Hosseiny F, Jetly R, Nicholson AA. Study protocol for a multi-session randomized sham-controlled trial of PCC- and amygdala-targeted neurofeedback for the treatment of PTSD. BMC Psychiatry. 2025 Jul 15;25(1):698. doi: 10.1186/s12888-025-07050-5. PMID 40665286